CLINICAL TRIAL: NCT01064167
Title: Tranexamic Acid Reduces Blood Loss After Off-pump Coronary Artery Bypass Grafting
Brief Title: Tranexamic Acid in Off-pump Coronary Surgery
Acronym: TAOPCAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Lihuan Li/Professor & Chief, Dep. of anesthesiology, Cardiovascular Institute and Fuwai Hospital, CAMS and PUMC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWMZ013
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Results first posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Off Pump Coronary Artery Bypass Surgery
Keywords: Tranexamic Acid; off-pump coronary Artery Bypass
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid group (Experimental)
  Interventions: Drug: Tranexamic Acid
- Control group (Placebo Comparator)
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — In tranexamic acid group, tranexamic acid, 1 g, was given 20 minutes before incision and 400 mg/h during the entire surgical procedure. The patients from control group were infused with normal saline as a placebo.

SUMMARY:
The aim of this prospective, randomized, double-blinded, placebo-controlled study was to evaluate the effects of tranexamic acid, a synthetic antifibrinolytic drug, on the postoperative bleeding and transfusion requirements in patients undergoing off-pump coronary artery bypass graphing (OPCAB) surgery.

DETAILED DESCRIPTION:
Cardiac surgical procedures account for a large amount of allogeneic transfusion. Although postoperative bleeding seems to be attenuated by the avoidance of cardiopulmonary bypass (CPB), hemorrhagic complications are not completely eliminated and the consequent need for allogeneic transfusions are still major problems after OPCAB.

Tranexamic acid, a synthetic antifibrinolytic drug, has been shown to reduce blood loss and transfusion requirements in cardiac surgery with CPB. About 30% of patients in OPCAB studies still receive a transfusion. A few small sample size studies concerned with the use of in OPCAB surgery, found that tranexamic acid appear to be effective in reducing postoperative bleeding, however, the results on transfusion requirements are still inconsistency. The purpose of this study was to evaluate the effects of tranexamic acid on the postoperative bleeding and transfusion requirements in a larger number of patients undergoing OPCAB surgery. In addition, the effect of tranexamic acid on mortality, morbidity and resource utilization was examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective offpump coronary artery bypass surgery

Exclusion Criteria:

* A history of bleeding disorders
* Active chronic hepatitis or cirrhosis
* Chronic renal insufficiency (serum creatinine > 2 mg/dL)
* Preoperative anemia (Hb < 10 g/dL)
* Previous cardiac surgery
* Myocardial infarction < 7 days before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lihuan Li, M.D, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, Beijing, China

REFERENCES:
- [Derived] Wang G, Xie G, Jiang T, Wang Y, Wang W, Ji H, Liu M, Chen L, Li L. Tranexamic acid reduces blood loss after off-pump coronary surgery: a prospective, randomized, double-blind, placebo-controlled study. Anesth Analg. 2012 Aug;115(2):239-43. doi: 10.1213/ANE.0b013e3182264a11. Epub 2011 Jul 7. PMID 21737704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2009 to December 2009, 378 consecutive patients in Fuwai hospital scheduled for elective OPCAB were enrolled in the study. 118 patients were excluded for randomizatin because not meeting inclusion criteria(n=29), Refused to participate(n=81),and surgery cancelled(n=8).
Pre-assignment Details: Of the 260 patients randomized, 130 were allocated to each group. 14 patients in tranexamic acid group and 15 in placebo group were withdrawn from the study for convert to on-pump surgery in course of surgery.
Groups:
- Tranexamic Acid Group: Tranexamic acid 1g was administered as a bolus injection 20 minutes before the incision and followed by a continuous infusion of 400 mg/h until the completion of the surgery.
- Control Group: The placebo consisted of an equivalent volume of saline solution.
Period: Overall Study
Arm/Group | Tranexamic Acid Group | Control Group
Started | 130 | 130
Completed | 116 | 115
Not Completed | 14 | 15
Not completed — Protocol Violation | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid Group | Control Group | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 89 | 175
  >=65 years | 44 | 41 | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.0) | 60 (8.5) | 60.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 16 | 42
  Male | 104 | 114 | 218
Region of Enrollment [Number; unit: participants]
  China | 130 | 130 | 260

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Required Allogenic Red Blood Cells Transfusion
Time Frame: 1month postoperative
Population: As predefined by study protocol,Fourteen patients in the tranexamic acid group and Fifteen in the placebo group were withdrawn from the study due to conversion to on-pump surgery during the course of surgery.
Measure: Number; unit: participants
Arm/Group | Tranexamic Acid Group | Control Group
Number analyzed (Participants) | 116 | 115
participants | 37 | 54
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Control Group; Given that the frequency of RBC transfusion for OPCAB surgery is about 55%, to detect 35% reduction in TA group, with power=o.8 and α=0.05, a group of 107 patients in each arm is required. We estimated a crossover rate of 20%. The final sample size for randomization purposes increased to a total of 260 patients. The Chi-square test was used to test the differences in categorical variables between both groups.If one or more cells had an expected count less than 5, Fisher's Exact Test was used; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Postoperative Chest Tube Drainage
Time Frame: 24h postoperative
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Tranexamic Acid Group | Control Group
Number analyzed (Participants) | 116 | 115
ml | 654 (224) | 891 (295)
Statistical Analysis 1: Comparison: Tranexamic Acid Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Tranexamic Acid Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/115
Other Adverse Events (participants affected / at risk) | 0/116 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes